CLINICAL TRIAL: NCT03232372
Title: The Marginal Bone Loss in Implants of External Connection Versus Internal Connection and Submerged Implants Versus Non-submerged Implants
Brief Title: The Marginal Bone Loss in Dental Implants
Acronym: BL-Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Natalia Palacios Garzón, PhD student (Universitat de Barcelona), University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUB
Record Dates: First submitted 2017-07-20; First posted 2017-07-28 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Dental Implants
Keywords: Bone loss, dental implant desing
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: To randomize we will use the application created by a computer programmer that generates random numbers.
  In each jaw, each edentulous space will be randomly assigned (A, B, C, D, ..). Following the alphabetical order to each letter will be assigned randomly the connection to use, as detailed below:
  * 2 edentulous spaces: A: c. External or c. Internal (random) B: the one that is pending (The type of internal connection (crestal or infracrestal) will be chosen at random.)
  * 3 edentulous spaces: A: c. External, c. Crestal or infracrestal internal B: randomly choose between the two remaining options C: the one that is pending
Who Masked: Participant
Masking Description: Blind study The RX examiner and the person performing the resonance frequency measurements would be independent of the surgeons who placed the implants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- External-Connection non-submerged Imp (Experimental): We will place implants with external connection and non- submerged to assess the bone loss around
  Interventions: Device: External-Connection non-submerged Imp
- Internal Connection Submerged implants (Experimental): We will place implants with internal connection and submerged to assess the bone loss around
  Interventions: Device: Internal Connection Submerged implants
- Internal Connection non-Submerged Impl (Experimental): We will place Internal connection implant and non-Submerged Implants to assess the bone loss around
  Interventions: Device: Internal Connection non-Submerged Impl

INTERVENTIONS:
Device: External-Connection non-submerged Imp — Through a surgical procedure, we will implant implant whit external connection and non submerged to patients.
  Arms: External-Connection non-submerged Imp
Device: Internal Connection Submerged implants — Through a surgical procedure, we will implant implant whit internal connection and submerged to patients.
  Arms: Internal Connection Submerged implants
Device: Internal Connection non-Submerged Impl — Through a surgical procedure, we will implant implant whit internal connection and non-submerged to patients.
  Arms: Internal Connection non-Submerged Impl

SUMMARY:
When an implant is placed, it is assumed that there will be a loss of bone in the more coronal area around it. The placement of the implant in relation to bone level, either crestal or subcrestal and the type of connection chosen, either external connection or internal connection, have been related as one of the factors that caused this loss. The preservation of the peri-implant bone influences the shape and contour of the underlying soft tissues, which are important for the aesthetic result of the treatment and for the success of the same.

Hypothesis: The hypothesis is that there are no differences between the external and internal connection with regard to marginal bone loss. In implants placed at the crestal and subcrestal level, the hypothesis is that there is greater marginal bone loss in implants placed at the subcrestal level.

Objectives: Main: To evaluate the marginal bone loss around implants of internal connection and external connection. Secondary: To compare the loss of bone in implants of internal connection placed at crestal and subcrestal level. To evaluate intra and post-operative complications.

Material and methods: A prospective and randomized radiological study will be performed. 150 implants will be placed in patients who must present partial edentulism and require the replacement of at least 2 crowns on implants in the same jaw. In a randomized manner, implants of external connection and internal connection will be placed. Other features such as surface treatment type of the implant will be similar in both types of implants to reduce bias.

With this study the investigators will try to define if there is a procedure in when to the connection of the implant and the location of this, that is more beneficial with respect to the preservation of bone.

DETAILED DESCRIPTION:
Implant dentistry has undergone major development and expansion since the nineteen sixties, when Dr. Branemark (Sweden) introduced the concept of osseointegration. The use of implants to replace missing teeth and restore function has presented a high success rate and long-term survival. For this reason rehabilitation by means of implants has become standard and well accepted by patients, who increasingly demand treatments offering greater comfort and aesthetics. Implant-based treatments must fulfill a range of physiological, functional and aesthetic criteria before they can be considered successful. These include osseointegration stability and duration, absence of pathological processes, and aesthetics that satisfy the patient.

There are diverse types of implants and corresponding systems that connect the implant to the prosthesis. Implant connections fall into two main groups: External and Internal Connection.

When an implant is placed, it is estimated that there will be bone loss around this during the first year, both horizontally and vertically. Actually is considered successful if the loss of crestal bone around the implant is less than 1.5mm during the first year and less than 0.2 annually in the next. This bone loss continues to occur despite the new designs of implants that try to stop it. The preservation of the peri-implant bone is an important factor for the success of the same. The quantity and quality influence the shape and contour of the overlying soft tissues, which are important for the aesthetic result of the treatment. The hypothesis is that there are no differences between the external and internal connection with regard to marginal bone loss. In implants placed at the crestal and subcrestal level, the hypothesis is that more marginal bone is loss in implants placed at the subcrestal level design.

A prospective randomized controlled, split-mouth clinical trial with a sample size of 50 implants per arm is proposed.

Population of the study Patients attended in HOUB (Hospital Odontológico Universitario de Bellvitge. Master of Medicine Surgery and Implantology and Master of Dentistry in Oncology and Immunocompromised Patients).

Inclusion criteria Patients of general age who present partial edentulism in the mandible and / or maxilla and require the replacement of at least 2 teeth by implants in the same maxilla. The teeth must have been removed at least 4-6 months before implant placement. The minimum required bone height would be 6mm, which would be determined by an orthopantomography (1: 1) to be performed in all cases. The space where the implants are placed should have sufficient bone volume that does not require regeneration (height> 6mm and bone width> 5mm). If expansion is to be done, it should be done in both techniques. The minimum distance from one implant to the adjacent teeth should be at least 1.5 mm, and in the case of two or more adjacent implants, at least 3 mm between them.

Intervention 150 implants will be placed (50 of external connection and 100 of internal connection: 50 with design for infracrestal placement and crestal-level.) Following the inclusion criteria, patients should require the replacement of at least two teeth in the same jaw.

To randomize we will use the application created by a computer programmer that generates random numbers.

All implants will be placed by the students of 3rd of Master, using the same surgical protocol.

Post-operative monitoring and follow-up visits Once the implants are placed, a period of osseointegration of 4 months will be left in the maxilla and 3 in the mandible. The control visits to assess clinical aspects were performed by the principal investigator at the following times: (0) prior to implant placement, (1) implant placement, (2) at 7 (+/- 1) days of placing the implant, where it will be used to remove the suture, (3) within 15 days (+/- 2 days) of placing the implant, (4) one month after placement, (5) 3 months (+/- 2 weeks) if it is placed in the mandible and at 4 months (+/- 2 weeks) in the jaw, when the healing pillar will be placed, (6) one week later, ) (+/- 1 day) at the printing press, (8) at 7 (+/- 1 day), where a metal test would be performed and (9) in the following week (+/- 1 Day), in the placement of the prosthesis, (10) 6 months after placement of the prosthesis and (11) 12 months after placement of the prosthesis.

The X-ray control, to compare bone loss, would be performed by an independent evaluator at the following times: (T1) prior to implant placement, (T2) on the day of implant placement, (T3) per month, (T4) at the time of placement of the implant Prosthesis (without specifying in which month), (T5) at 6 months after loading and (T6) one year after occlusal loading.

The stability implants, would be performed by an independent evaluator using the analysis of the resonance frequency (Penguin device) The measurements will be made the day of implant placement, the day of placement of the healing abutment (two-three months after implant placement) and the day of delivery of the crown (3-4 months after placement of the implant)

Study variables - Primary study variables: Percentage of bone loss

- Secondary study variables: Tobacco consumption Plate Index (PLI) Bleeding index (SBI) Implant stability ratio (ISQ) Intra and postoperative parameters

Statistic analysis The data will be entered into an Excel database and processed using the statistical package (SPSS )Windows. The level of statistical significance will be p <0.05.

A descriptive study of all the variables and the relationship between bone loss and the implant system or the different variables will be analyzed by the t-student for the independent data or by non-parametric tests (Mann-W-U ) If the distribution is not normal.

The Chi-squared test will be used to analyze the qualitative variables. Multiple regression analysis will be used to evaluate the association between the dependent variable (bone loss at 0, 1, 4, 6 and 12 months) and the independent variables, internal connection or external connection. All the variables that could potentially affect the study relationship, such as age, sex, smoking, and oral hygiene, were used as control variables in the regression.

Blind study

Ethical aspects The study would be carried out in accordance with the general recommendations of the 1964 Declaration of Helsinki for biomedical research in humans.

Eligible patients would be explained in detail to the study protocol and given an information sheet to those who enroll, they would be given to sign two informed consents; The first, explaining the risk and complications derived from implant placement surgery and the second where they agree to participate in the study. All patients will have a medical history and a data collection sheet attached to their history

ELIGIBILITY:
Inclusion Criteria:

* Patients of general age who present partial edentulism in the mandible and / or maxilla and require the replacement of at least 2 teeth by implants in the same maxilla.
* The teeth must have been removed at least 4-6 months before implant placement.
* The minimum required bone height would be 6mm, which would be determined by an orthopantomography (1: 1)

Exclusion Criteria:

* History of use of bisphosphonates
* Evidence of serious systemic diseases such as recent infarction
* Uncontrolled diabetes, coagulation disorders, cancer, psychiatric contraindications,
* Active infection in the area of the implants
* Absence of an antagonist in the area of implant placement
* Pharmacological treatments capable of affecting gingival health
* Pregnant or lactating women.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-05-08 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2022-02-17 (Estimated)

PRIMARY OUTCOMES:
A COMPARISON BETWEEN THE DIFFERENT CONNECTIONS AND POSITIONING OF THE IMPLANTS REGARDING THE BONE OF LOSS | 1,4 years around
  By means of measurements in millimeters in the radiographs, the loss of bone will be compared. These measurements will be made one month after the placement of the implant, at 3-4 months in the placement of the crown, 6 months after placement of the crown and one year after placement of the crown

OTHER OUTCOMES:
ANALYSIS OF THE RESONANCE FREQUENCY | 4-5months around
  Using the Penguin device, the investigators measure the coefficient of stability of the implant. Measurements will be made the day of implant placement, the day of placement of the healing abutment (two-three months after implant placement) and the day of delivery of the crown (3-4 months after placement Of the implant)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Palacios Garzón, PhD student, Principal Investigator — HUBellvitge Recruiting; José López López, PhD, Study Director — Hospital Universitari de Bellvitge
Locations (1):
- Natalia Palacios Garzon, Barcelona, Spain

REFERENCES:
- [Background] Pozzi A, Tallarico M, Moy PK. Three-year post-loading results of a randomised, controlled, split-mouth trial comparing implants with different prosthetic interfaces and design in partially posterior edentulous mandibles. Eur J Oral Implantol. 2014 Spring;7(1):47-61. PMID 24892113
- [Background] Penarrocha-Diago MA, Flichy-Fernandez AJ, Alonso-Gonzalez R, Penarrocha-Oltra D, Balaguer-Martinez J, Penarrocha-Diago M. Influence of implant neck design and implant-abutment connection type on peri-implant health. Radiological study. Clin Oral Implants Res. 2013 Nov;24(11):1192-200. doi: 10.1111/j.1600-0501.2012.02562.x. Epub 2012 Aug 28. PMID 22925048
- [Background] Galindo-Moreno P, Fernandez-Jimenez A, O'Valle F, Monje A, Silvestre FJ, Juodzbalys G, Sanchez-Fernandez E, Catena A. Influence of the crown-implant connection on the preservation of peri-implant bone: a retrospective multifactorial analysis. Int J Oral Maxillofac Implants. 2015 Mar-Apr;30(2):384-90. doi: 10.11607/jomi.3804. PMID 25830399